CLINICAL TRIAL: NCT03655106
Title: Standard vs Long IV Catheter Long-Term IV Survival Comparison
Brief Title: Ultrasound Guided Catheter Length Survivability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Amit Bahl, Director of Emergency Ultrasound, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-185
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Catheter Complications
Keywords: Ultrasound guided intravenous access; vascular access; extended dwell catheter; IV survival
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Intervention Model Description: Randomized control parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Long IV 4.78 cm 20 g catheter (Active Comparator): Placement of Standard Long IV 4.78 cm 20 g catheter
  Interventions: Device: Standard Long IV 4.78 cm 20 g catheter
- Ultra-Long IV 6.35 cm 20 g catheter (Experimental): Placement of Ultra-Long length IV 6.35 cm 20 g catheter
  Interventions: Device: Ultra-Long IV 6.35 cm 20 g catheter

INTERVENTIONS:
Device: Standard Long IV 4.78 cm 20 g catheter — Standard Long IV 4.78 cm 20 g catheter
  Arms: Standard Long IV 4.78 cm 20 g catheter
Device: Ultra-Long IV 6.35 cm 20 g catheter — Ultra-Long IV 6.35 cm 20 g catheter
  Arms: Ultra-Long IV 6.35 cm 20 g catheter

SUMMARY:
In patients with difficult IV access, ultrasound-guided catheter insertion is a preferred technique. However, many peripheral catheters fail and must be replaced, adding extra pain and difficulty for the patient, and requiring more healthcare provider time to maintain. In preliminary studies, we determined that catheters which extend further into the vein have a smaller failure rate. This study will compare two lengths of catheters to see if the longer catheters have better survival in a population of patients who have difficult IV access. Patients will be randomized to receive a standard length or extra-long venous catheter, which will be monitored daily for functionality during the patient's hospital course.

DETAILED DESCRIPTION:
Patients with poor intravenous (IV) access present a daily challenge to emergency department (ED) practitioners. Placement of an ultrasound (US)-guided peripheral IV catheter in this patient population is a viable and safe option. Ultrasound-guided IVs are often the last recourse for IV access before resorting to more invasive procedures in patients with difficult access. Successful cannulation with US-guided IV occurs in more than 90% of cases compared with 25-35% with traditional IV placement in patients with difficult vascular access. Once cannulated, however, the failure rate of IV catheters placed under ultrasound guidance is concerning compared with traditional blind IV placement. Overall failure rates after successful IV cannulation for US-guided IVs is 45-56% when compared to traditional IV placement which is 19-25%. Because failure rate is high, it is important to approach insertions methodically to improve survival rates. A variable that may alter the survival of US-guided IVs that has not been studied is the length of catheter that resides in the vein. Currently the general accepted rule is that an "adequate" amount of the catheter should be in the vein to avoid failure of the catheter. Our preliminary data focused on defining this relationship. In our study, 100% of catheters failed in which less than 30% of the catheter was placed within the vein and no failures in those IVs in which at least 65% of the catheter was in the vein. This study was performed by the PI at Beaumont this past year and is published in Emergency Medicine Journal.

This study is a prospective randomized controlled study of catheter longevity comparing a 4.78 cm (1.88 in) catheter to a longer 6.35 cm (2.5 in) catheter. Subjects will consist of a convenience sample of patients with difficult IV access presenting to the Beaumont Hospitals emergency department that require US-guided IV access.

Standard of care is defined as use of a readily available 1.88 inch IV catheter that is used daily by emergency department personnel. Following consent, patients will be randomized to the control arm using the standard 4.78 cm catheter, or the experimental arm using a 6.35 cm catheter. All catheters are 20 gauge in diameter.

After patient enrollment, the insertion tech, nurse or physician who has been credentialed in ultrasound-guided vascular access will place catheters in study subjects. Staff are expected to attempt a minimum of 3 attempts before enlisting another provider for help.

After initial assessment, follow-up functionality of the catheter will be assessed every 24 hours by the research team as long as the patient is hospitalized, up to 30 days. Function of the catheter will be assessed daily by research staff. Function is defined by a catheter's ability to draw back 5 ml of blood, flush with 5 ml normal saline without resistance, or if IV fluids or medication are continually infusing through the IV.

Other data variables collected include: patient pertinent medical history, vitals, age, sex, cannulation success or failure, vein diameter, length of catheter in vein as well as % length of the catheter in the vein, angle of insertion, number of venous access attempts, time to IV insertion (tourniquet to tegaderm), location of IV insertion, medications infused or use for ionic contrast injection for computed tomography.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Self-reported difficult IV Access Patient and any one of the following:

* Greater than 2 sticks in previous admission/hospital encounter
* History of rescue vascular access device (such as US-guided IV, PICC line, midline, or CVC)
* End-stage renal disease on dialysis
* History of IV Drug Use
* History of Sickle Cell Disease

Exclusion Criteria:

Age under 18 years old

* Voluntary withdrawal or refusal to participate
* Previous enrollment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD, Principal Investigator — Director of Emergency Ultrasound
Locations (1):
- Beaumont Hospitals, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahl A, Hijazi M, Chen NW, Lachapelle-Clavette L, Price J. Ultralong Versus Standard Long Peripheral Intravenous Catheters: A Randomized Controlled Trial of Ultrasonographically Guided Catheter Survival. Ann Emerg Med. 2020 Aug;76(2):134-142. doi: 10.1016/j.annemergmed.2019.11.013. Epub 2020 Jan 16. PMID 31955940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Long IV 4.78 cm 20 g Catheter | Ultra-Long IV 6.35 cm 20 g Catheter
Started | 135 | 135
Completed | 126 | 131
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Duplicate Enrollment | 1 | 1
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Long IV 4.78 cm 20 g Catheter | Ultra-Long IV 6.35 cm 20 g Catheter | Total
Number analyzed (Participants) | 126 | 131 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (18.6) | 60.2 (18.2) | 59.2 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 92 | 184
  Male | 34 | 39 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 126 | 131 | 257

OUTCOME MEASURES:

1. Primary Outcome: Duration of IV Survival
Description: Function is defined by a catheter's ability to draw back 5 ml of blood, flush with 5 ml normal saline without resistance, or if IV fluids or medication are continually infusing through the IV. Function is assessed daily by research staff.
Time Frame: 30 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Standard Long IV 4.78 cm 20 g Catheter | Ultra-Long IV 6.35 cm 20 g Catheter
Number analyzed (Participants) | 126 | 131
hours | 92 [71 to 120] | 136 [116 to 311]

2. Secondary Outcome: Thrombosis
Description: Number of patient with thrombosis upper extremity superficial or deep venous thrombosis as measured by venous doppler study in symptomatic patients
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Long IV 4.78 cm 20 g Catheter | Ultra-Long IV 6.35 cm 20 g Catheter
Number analyzed (Participants) | 126 | 131
Participants | 0 | 0

3. Secondary Outcome: Infection
Description: Number of patient with infection as defined as the patient meeting the laboratory-confirmed bloodstream infection criteria as defined by the Centers for Disease Control.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Long IV 4.78 cm 20 g Catheter | Ultra-Long IV 6.35 cm 20 g Catheter
Number analyzed (Participants) | 126 | 131
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 Days post IV catheter insertion
Description: Thrombosis was assessed based on upper extremity venous duplex results in symptomatic patients.
  Catheter related bloodstream infection was determined by the institutional Department of Epidemiology based on the definition of catheter related bloodstream infection provided by the Centers of Disease Control.
Arm/Group | Standard Long IV 4.78 cm 20 g Catheter | Ultra-Long IV 6.35 cm 20 g Catheter
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/131
Other Adverse Events (participants affected / at risk) | 0/126 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT03655106/Prot_SAP_000.pdf